CLINICAL TRIAL: NCT02524535
Title: Alliance With Therapeutic Entourage in Support of Young Suicidal
Acronym: IPSI2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 06-088
Record Dates: First submitted 2015-08-13; First posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide | interventions — Therapeutic Alliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Therapetic alliance (Other)
  Interventions: Other: Therapeutic alliance

INTERVENTIONS:
Other: Therapeutic alliance

SUMMARY:
Regardless of age, the quality of hospital care, the confidence that the young can have in the health care team, joining parents are pivotal elements and influence followed. Family support is all the more important as 14% of young people realize a new suicidal act within three months of hospitalization for attempted suicide, and that the essential predictors appear to be the young age and quality of intra-family relationships.

The main objective of this study is to determine, through the construction of an instrument to quantify the therapeutic alliance, defined by the characteristics of the mobilization of the entourage and the mutual commitments in the care of nursing teams and the entourage, the role of early therapeutic alliance with the entourage of suicidal youth 13-40 years, whether primosuicidants or repeat offenders, on short and medium term recurrences and early mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 13-40 years
* From male or female
* Supported the waning of a suicidal gesture.
* speaking and writing fluent French
* living in Upper or Lower Normandy
* signed informed consent form, and at least one of his parents after oral and written information about the study for minors.

Exclusion Criteria:

* Age <13 years or > 40 years
* Do not live in the Upper and Lower Normandy regions
* Detained patient
* forced hospitalization
* Patient under guardianship
* Patient with severe somatic pathology (cancer, heart failure, kidney or respiratory, central neurological disorder), scalable, or likely to be life-threatening within a period of less than one year
* Refusal to participate in the study
* Inability to respond

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 292 (Actual)
Dates: Start 2007-04; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
characteristics of the mobilization of the entourage evaluated with Family Assessment Device | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- service de pédopsychiatrie, CHU de Caen, Caen, France